CLINICAL TRIAL: NCT04642027
Title: PSMA-PET Guided Hypofractionated Salvage Prostate Bed Radiotherapy of Biochemical Failure After Radical Prostatectomy for Prostate Cancer
Brief Title: PSMA-PET Guided Hypofractionated Salvage Prostate Bed Radiotherapy
Acronym: PERYTON
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT2020-01
Record Dates: First submitted 2020-08-13; First posted 2020-11-24 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer; Cancer Recurrence
Keywords: PSMA-PET/CT; Salvage; Hypofractionation; Radiotherapy; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: 2 randomised arms
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): Conventional sEBRT
  Interventions: Radiation: Conventional sEBRT
- Hypofractionation (Experimental): Hypofractionated sEBRT
  Interventions: Radiation: Hypofractionated sEBRT

INTERVENTIONS:
Radiation: Conventional sEBRT — A total dose of70 Gy in 35 daily fractions of 2 Gy during 7 weeks
  Other Names: Conventional salvage external beam radiation therapy
  Arms: Conventional
Radiation: Hypofractionated sEBRT — A total dose of 60 Gy in 20 daily fractions of 3 Gy during 4 weeks
  Other Names: Hypofractionated salvage external beam radiation therapy
  Arms: Hypofractionation

SUMMARY:
After radical prostatectomy approximately 15-40% of men develop a biochemical recurrence (BR) within 5 years.

The standard treatment of post-prostatectomy BR is salvage external beam radiation therapy (sEBRT). sEBRT can provide long-term disease control; with 5 year biochemical progression-free survival (bPFS) up to 60% and with most treatment failures in the first 2 years after sEBRT.

The main goal of this project is to investigate whether the oncologic outcome in patients with post-prostatectomy recurrent PCa can be improved, by increasing the biological effective radiation dose using a hypofractionated schedule of 20 x 3 = 60 Gy.

The study is designed as a prospective open phase III randomized multicenter trial. All patients with biochemical recurrence with a PSA < 1.0 ng/ml after radical prostatectomy for prostate cancer without evidence of lymph nodes or distance metastases will be included. PSA progression after prostatectomy defined as two consecutive rises with the final PSA > 0.1 ng/mL or three consecutive rises will be included.

All eligible patients will be randomized to one of the following two treatment arms:

Arm 1 = Conventional sEBRT to apply a total dose of 70 Gy in 35 daily fractions of 2 Gy during 7 weeks.

Arm 2 = Hypofractionated sEBRT to apply a total dose of 60 Gy in 20 fractions of 3 Gy during 4 weeks.

The primary endpoint will be the 5-year progression-free survival (PFS) after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prostate adenocarcinoma treated with radical prostatectomy;
* Tumour stage pT2-4, R0-1, pN0, or cN0, cNx according to the UICC TNM 2009, only with Gleason score available;
* No lymph node or distant metastases. A recent PSMA-PET scan (< 60 days) without evidence of lymph node or distant metastases;
* PSA progression after prostatectomy defined as two consecutive rises with the final PSA > 0.1 ng/mL or 3 consecutive rises. The first value must be measured at least 6 weeks after radical prostatectomy;
* PSA at inclusion < 1.0 ng/mL;
* WHO performance status 0-2 at inclusion;
* Age at inclusion between 18 and 80 years;
* Written (signed and dated) informed consent prior to registration.

Exclusion Criteria:

* Prior pelvic irradiation, (chemo)hormonal therapy or orchiectomy;
* Previous or concurrent active invasive cancers other than superficial non-melanoma skin cancers;
* Patients with positive nodes or with distant metastases based on the surgical specimen of lymphadenectomy or the following minimum diagnostic workup: PSMA-PET/CT scan, 60 days prior to registration;
* Double-sided metallic hip prosthesis;
* Inability or unwillingness to understand the information on trial-related topics, to give informed consent or to fill out QoL questionnaires.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 538 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
5-year progression-free survival | 5 years
  Defined as biochemical progression, clinical progression, loco-regional or distant progression or start with hormonal therapy, whichever occurs first

SECONDARY OUTCOMES:
Acute grade ≥ 2 gastrointestinal toxicity | Up to 3 months after completion of the RT
  As assessed using physician-reported score: Common Terminology Criteria for adverse events version 5.0 (CTCAE-5) toxicity score with a scale of 1 - 4.
Acute grade ≥ 2 genitourinary toxicities | Up to 3 months after completion of the RT
  As assessed using physician-reported score using questionnaires (CTCAE 5.0 toxicity score).
Late grade ≥ 2 gastrointestinal toxicity | Up to 5 years after completion of the RT
  As assessed using physician-reported score (CTCAE 5.0 toxicity score).
Late grade ≥ 2 genitourinary toxicity | Up to 5 years after completion of the RT
  Using physician-reported score (CTCAE 5.0 toxicity score).
Quality of life after radiation | Up to 5 years after completion of the RT
  As assessed using patient-reported questionnaires: measurend with European platform of cancer research-QLQ C30
Metastasis-free survival | 5 years
  Time from randomisation to the date of metastases reported by CT scan, MRI scan or PSMA-PET/CT during the follow up (date scan).
Prostate cancer-specific mortality | 5 years
  Prostate cancer-specific mortality.
Overall survival | 5 years
  Overall survival
Acute grade ≥ 2 gastrointestinal toxicity | Up to 3 months after completion of the RT
  Using patient-reported questionnaires (Radiation Therapy Oncology Group (RTOG) / European platform of cancer research (EORTC) toxicity questionnaires with grade 1 to 4).
Acute grade ≥ 2 genitourinary toxicities | Up to 3 months after completion of the RT
  Using patient-reported questionnaires (Radiation Therapy Oncology Group (RTOG) / European platform of cancer research (EORTC) toxicity questionnaires with grade 1 to 4).
Late grade ≥ 2 genitourinary toxicity | Up to 5 years after completion of the RT
  Using patient-reported questionnaires (Radiation Therapy Oncology Group (RTOG) / European platform of cancer research (EORTC) toxicity questionnaires with grade 1 to 4).
Quality of life after radiation | Up to 5 years after completion of the RT
  As assessed using patient reported quatinnaires: European platform of cancer research-Quality of Life Questionnaire - Prostate Cancer Module (PR 25).

CONTACTS AND LOCATIONS:
Overall Officials: S. Aluwini, Dr., Principal Investigator — University Medical Center Groningen
Locations (13):
- Netherlands (13):
  - Radiotherapiegroep, Arnhem, Gelderland
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Maastro Clinic, Maastricht, Limburg
  - Catharina-Hospital, Eindhoven, North Brabant
  - Verbeeten Institute, Tilburg, North Brabant
  - Amsterdam UMC (Location VUmc), Amsterdam, North Holland
  - Radiotherapiegroep, Deventer, Overijssel
  - Radiotherapy Institute Friesland, Leeuwarden, Provincie Friesland
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Haga Hospital, The Hague, South Holland
  - Zuidwest Radiotherapeutisch Instituut (ZRTI), Flushing
  - UMCG, Groningen

REFERENCES:
- [Derived] Staal FHE, Janssen J, Brouwer CL, Langendijk JA, Ng Wei Siang K, Schuit E, de Jong IJ, Verzijlbergen JF, Smeenk RJ, Aluwini S. Phase III randomised controlled trial on PSMA PET/CT guided hypofractionated salvage prostate bed radiotherapy of biochemical failure after radical prostatectomy for prostate cancer (PERYTON-trial): study protocol. BMC Cancer. 2022 Apr 15;22(1):416. doi: 10.1186/s12885-022-09493-5. PMID 35428210